CLINICAL TRIAL: NCT03565107
Title: Characterization of Methylation Pattern in Human Germ Cells of Patients with the Desire to Have Children Undergoing Intracytoplasmic Sperm Injection Treatment
Brief Title: Characterization of Methylation Pattern in Human Germ Cells of Patients Undergoing ICSI Treatment
Status: Completed | Type: Observational
Sponsor: Infertility Treatment Center Dortmund (Other)
Collaborators: University of Wuerzburg (Other)
Responsible Party: Sponsor
Other Study IDs: Methylation in Germ cells
Record Dates: First submitted 2018-06-05; First posted 2018-06-21 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Female Infertility; Gene Deregulation
Keywords: Epigenetic; Female age; Gene regulation; Methylation pattern
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Immature oocytes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Female Patients: ICSI treatment because of male subfertility

SUMMARY:
There is increasing evidence that exposure to environmental factors in early development is associated with an increased risk of metabolic and other common diseases. These increased disease risks are likely due to environmental-induced epigenetic changes leading to dysregulation of genes and signaling cascades. The best studied epigenetic modification in this context is DNA methylation. Preliminary studies have already shown that an increased father age or intracytoplasmic sperm injection affects methylation pattern in sperm or umbilical cord blood of children. Unlike sperm, less is known about the methylation of human oocytes and their susceptibility to environmental factors. The aim of this study is to analyze the methylation pattern of immature oocytes of women with decreased fertility. Based on the results of a large number of oocytes from different women, risk assessments could be made for individual factors such as the age of the patient, as well as correlations between the occurrence of changes in gene expression and the unfulfilled desire to have children. In addition, the methylation patterns in sperm from 20 patients are to be examined as reference patterns.

DETAILED DESCRIPTION:
Although more than five million children have been conceived worldwide through Assisted Reproduction Techniques (ARTs), little is known about potential effects of ART in later life. So far, the focus of reproductive research is based on the success rate of infertility treatment. There is increasing evidence that exposure to environmental substances, age of the patient or in vitro culture conditions in early development is associated with a life-long increased risk of metabolic and other common diseases. These increased disease risks are likely due to environmental-induced epigenetic changes leading to dysregulation of genes and signaling cascades. These include Beckwith-Wiedemann and Angelman syndrome.

The best studied epigenetic modification in this context is DNA methylation, which regulates the gene expression in a temporally and highly coordinated manner. Preliminary studies have already shown that an increased father age influences the pattern of methylation in the sperm and umbilical cord blood of children. Moreover, intracytoplasmic sperm injection (ICSI) also leaves epigenetic signatures in umbilical cord blood. Unlike sperm, little is known about the methylation of human oocytes and their susceptibility to environmental factors. The main reason for this is the difficulty of collecting human oocytes in sufficient numbers for genome-wide analysis. The aim of this study is to analyze the methylation pattern of immature oocytes, which are not suitable for further ICSI treatment, of women with decreased fertility. The products of gene expression and also the methylation of the DNA itself can be investigated using newly developed DNA sequencing methods. Based on the results of a large number of oocytes from different women, risk assessments could be made for individual factors such as the age of the patient, as well as correlations between the occurrence of changes in gene expression and the unfulfilled desire to have children. In addition, the methylation patterns in sperms from 20 patients are to be examined as reference.

ELIGIBILITY:
Inclusion Criteria:

- healthy females without sterility factors

Exclusion Criteria:

* Endometriosis
* Polycystic ovary syndrome (PCO)
* Neoplasia (ovary, Uterus, breast)
* Anti-Müllerian hormone (AMH) <1 ng/ml

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: female patients seeking ICSI treatment because of male subfertility
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Methylation pattern | 1 day (Directly after oocyte pick-up)
  Analysis of methylation pattern in immature oocytes (not suitable for further ICSI treatment). Methylation will be pointed out as number of methylated gene loci in comparison to the overall amount of analyzed gene loci.
Gene expression | 1 day (Directly after oocyte pick-up)
  Analysis of gene expression in immature oocytes (not suitable for further ICSI treatment) will be done by quantification of selected gene transcripts (in picogram).

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Dieterle, MD, Principal Investigator — Infertility Treatment Center Dortmund
Locations (1):
- Infertility treatment center Dortmund, Dortmund, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No